CLINICAL TRIAL: NCT03137134
Title: A Phase 1, Open-label, Single Dose Study To Evaluate The Effects Of Food And The Proton Pump Inhibitor, Esomeprazole, On The Pharmacokinetics Of Crizotinib In A Coated Microsphere Formulation In Adult Healthy Volunteers
Brief Title: A Study to Evaluate the Effects of Food and Esomeprazole on the Pharmacokinetics of Crizotinib in a Coated Microsphere Formulation.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A8081066; PPI/FE (Other: Alias Study Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-02 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Crizotinib; Esomeprazole

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Treatment A (Active Comparator): (reference) Crizotinib cMS 300 mg in fasted state
  Interventions: Drug: Crizotinib
- Treatment B (Experimental): (test) Crizotinib cMS 300 mg in fed state
  Interventions: Drug: Crizotinib
- Treatment C (Experimental): (test) 5 days of esomeprazole 40 mg followed by crizotinib cMS 300 mg in fasted state
  Interventions: Drug: Crizotinib; Drug: Esomeprazole
- Treatment D (Experimental): (test) 5 days of esomeprazole 40 mg followed by crizotinib cMS 300 mg with apple sauce.
  Interventions: Drug: Crizotinib; Drug: Esomeprazole
- Treatment E (Experimental): (test) 5 days of esomeprazole 40 mg followed by crizotinib cMS 300 mg with orange juice
  Interventions: Drug: Crizotinib; Drug: Esomeprazole

INTERVENTIONS:
Drug: Crizotinib — Crizotinib in a coated microsphere formulation
Drug: Esomeprazole — Proton pump inhibitor, esomeprazole
  Arms: Treatment C; Treatment D; Treatment E

SUMMARY:
This study will estimate the effect of food and the proton pump inhibitor, esomeprazole on the pharmacokinetics of crizotinib in a coated microsphere formulation.

DETAILED DESCRIPTION:
This study is an open-label, randomized, 4-period, 5-treatment, 6-sequence study in adult healthy volunteers. Subjects will receive up to four separate single oral 300 mg doses of a coated microsphere (cMS) formulation of crizotinib. Period 1 through Period 3 will evaluate the effect of food, and, the effect of multiple doses of a gastrointestinal acid reducing agent, esomeprazole, in fasted state, on the pharmacokinetics (PK) of crizotinib cMS. Period 4 will evaluate whether apple sauce or orange juice may reduce the effect of multiple doses of esomeprazole on the PK of crizotinib cMS, if there is an effect.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects and female subjects of nonchildbearing potential between 18 and 55 years old.
2. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug test.
4. Subjects who currently smoke.
5. History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
6. Subjects with history of known sensitivity to esomeprazole or substituted benzimidazoles.
7. Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study drug.
8. Screening supine BP greater than or equal to 140 mm Hg (systolic) or greater than or equal to 90 mm Hg (diastolic), following at least 5 minutes of supine rest.
9. Screening supine 12-lead triplicate ECG demonstrating a corrected time from the beginning of the Q wave to the end of the T wave corresponding to electrical systole (QTc) interval >450 msec or a QRS complex >120 msec.
10. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    1. Aspartate aminotransferase (AST) or ALT level greater than or equal to 1.5 × upper limit of normal (ULN);
    2. Total bilirubin (TBili) level greater than or equal to 1.5 × ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is less than or equal to ULN.
11. Male subjects who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product.
12. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of IP.
13. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
14. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
15. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
16. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
17. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or crizotinib cMS and/or esomeprazole administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Crizotinib pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours post-dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | Crizotinib pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours post-dose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Maximum Observed Plasma Concentration (Cmax) | Crizotinib pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours post-dose

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Crizotinib pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours post-dose
Time of last observed concentration (Tlast) | Crizotinib pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours post-dose
Plasma Decay Half-Life (t1/2) | Crizotinib pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | Crizotinib pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | Crizotinib pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 35 calendar days after the last crizotinib dose
Number of Participants With Abnormal Electrocardiogram (ECG) | Baseline up to 35 calendar days after the last crizotinib dose
Number of Adverse Events by Severity | Baseline up to 35 calendar days after the last crizotnib dose
  An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs are classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081066&StudyName=A+Phase+1%2C+Open-label%2C+Single+Dose+Study+To+Evaluate+The+Effects+Of+Food+And+The+Proton+Pump+Inhibitor%2C+Esomeprazole%2C+On+The+Pharmacokinetics+Of+Crizotinib+In+A+Coated+Microsphere+Formulation+In+Adult+Healthy+Volunteers